CLINICAL TRIAL: NCT03348189
Title: SpO2 Hypoxia Accuracy Validation Study
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP3093
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: US Export: Yes

GROUPS / COHORTS (1):
- Observational: Healthy males and females
  Interventions: Other: Pulse Oximeter

INTERVENTIONS:
Other: Pulse Oximeter — Pulse Oximeter

SUMMARY:
The primary objective of this study is to evaluate the % oxygen saturation by pulse oximetry accuracy of a combined pulse oximetry system which consists of a Nonin sensor ), an adaptor cable, and an oximetry system during non-motion conditions.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the %SpO2 accuracy of a combined pulse oximetry system which consists of a Nonin sensor ), an adaptor cable, and an oximetry system during non-motion conditions.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female
* The subject is of any racial or ethnic group
* The subject is ≥ 30 kg (≥ 66 pounds) in weight (self-reported)
* The subject has at least one finger height of 0.2 - 1.0 inch (based on measurement)
* The subject is between 18 years and 50 years of age (self-reported)
* The subject shows no evidence of medical problems as indicated by satisfactory completion of the health assessment form
* The subject has given written informed consent to participate in the study
* The subject is both willing and able to comply with study procedures.

Exclusion Criteria:

* The subject has a BMI greater than 31 (based on weight and height)
* The subject has had any relevant injury at the sensor location site (self-reported)
* The subject has deformities or abnormalities that may prevent proper application of the device under test (based on examination)
* The subject is current smoker (self-reported)
* The subject has a known respiratory condition (self-reported)
* The subject has a known heart or cardiovascular condition (self-reported)
* The subject is currently pregnant, is actively trying to get pregnant, or who has a positive urine pregnancy test on the day of the study
* The subject has a clotting disorder (self-reported)
* The subject has Raynaud's Disease (self-reported)
* The subject is known to have a hemoglobinopathy (self-reported)
* The subject is on blood thinners or medication with aspirin (self-reported)
* The subject has unacceptable collateral circulation from the ulnar artery (based on examination)
* The subject is unwilling or unable to provide written informed consent to participate in the study
* The subject is unwilling or unable to comply with the study procedures
* The subject has another health condition which in the opinion of the principal investigator makes him/her unsuitable for testing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A minimum of 12 subjects will be enrolled. The subject population will include both male and female subjects with a variety of skin tones.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
SpO2 Hypoxia Accuracy Validation Study | Through study completion, 3 months average
  Values from the test device will be compared to the values from co-oximetry to determine accuracy of the test device.

CONTACTS AND LOCATIONS:
Overall Officials: Dena Raley, Study Director — Clinimark, LLC
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No